CLINICAL TRIAL: NCT06077253
Title: Danish Angle Closure Prevention Trial
Acronym: DAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DAP
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Primary Angle Glaucoma Closure Suspect

STUDY DESIGN:
Intervention Model Description: One eye intervention (prophylactic iridotomy), one eye no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): One eye iridotomy, contralateral eye no intervention
  Interventions: Procedure: Iridotomy

INTERVENTIONS:
Procedure: Iridotomy — Peripheral iridotomy (size >200µm)

SUMMARY:
To determine whether primary angle closure suspects (PACS) in a Caucasian population benefit from prophylactic laser iridotomy.

DETAILED DESCRIPTION:
Prospective, randomised paired-eye design clinical trial comparing peripheral laser iridotomy in one eye with observation in the other over 5-years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary angle closure suspect: ≥180 degrees (cumulative) irido-trabecular contact on darkroom gonioscopy, IOP<21mmHg, no peripheral anterior synechiae, no glaucomatous optic neuropathy
* Best-corrected visual acuity (BCVA) >0.8 on both eyes
* Caucasian

Exclusion Criteria:

* Pseudophakia
* Previous iridotomy
* Clinically significant cataract with indication for surgery,
* Gaucoma
* Uveitis
* Unstable retinal conditions
* Ocular malignancies
* PEX
* PDS
* Systemic or ocular corticosteroid treatment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 5 year
  GAT: ≥24mmHg or ≥22mmHg on two separate occasions
Glaucoma | 5 year
  The presence of glaucomatous optic neuropathy with visual field loss compatible with glaucoma. Glaucomatous optic neuropathy defined as loss of neuroretinal rim (notch or erosion), a vertical cup-to-disc ratio of more than 0.7, nerve fiber layer defect attributable to glaucoma, or both.
Acute Primary Angle Closure | 5 year
  Presence of at least 2 of the following symptoms: ocular or periocular pain; nausea, vomiting, or both; an antecedent history of intermittent blurring of vision with haloes and IOP of more than 30 mmHg and presence of at least 3 of the following signs: conjunctival injection, corneal epithelial edema, mid-dilated unreactive pupil, glaukomflecken, and shallow anterior chamber;

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Telinius, Principal Investigator — Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Odense University Hospital, Odense
  - Sygehus Lillebælt, Vejle